CLINICAL TRIAL: NCT05252923
Title: Endothelial Protection in Convalescent COVID-19 Patients. The Effect of Sulodexide on Serum Levels of Biomarkers for Endothelial Dysfunction. A Pilot Prospective, Randomized, Open-label, Investigator-initiated Trial.
Brief Title: Endothelial Protection in Convalescent COVID-19 Patients
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Lack of the eligible patients
Sponsor: Pirogov Russian National Research Medical University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: SDXbioCOVID-19
Record Dates: First submitted 2022-02-21; First posted 2022-02-23 (Actual); Last update posted 2025-06-13 (Actual); Status verified 2025-01

CONDITIONS: Endothelial Dysfunction; Inflammation; Thrombosis; COVID-19
MeSH Terms: conditions — Inflammation; Thrombosis; COVID-19 | interventions — glucuronyl glucosamine glycan sulfate

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sulodexide (Experimental): Standard treatment plus oral sulodexide
  Interventions: Drug: Sulodexide
- Control (No Intervention): Standard treatment only

INTERVENTIONS:
Drug: Sulodexide — Sulodexide 250 LSU 1 oral capsule twice daily for 8 weeks
  Arms: Sulodexide

SUMMARY:
This pilot open-label randomized controlled trial aims to assess if treatment with sulodexide may improve the endothelial status and inflammatory response in post-COVID-19 patients. Survived inpatients with severe-to-critical COVID-19 within 14 days after discharge are randomized to receive sulodexide 250 LSU 1 oral capsule twice daily or no treatment for 8 weeks. Biomarkers of endothelial dysfunction, inflammation, and prothrombotic changes are assessed at 0, 4, and 8 weeks. The hypothesis is that affected endothelial function, pro-inflammatory, and pro-thrombotic changes could be improved with sulodexide treatment in convalescent COVID-19 patients who suffered a severe-to-critical clinical presentation and have chronic comorbidities of high risk for endothelial dysfunction.

ELIGIBILITY:
Inclusion Criteria:

* over 18 years old
* male or female
* documented PCR SARS-CoV-2 positive test
* COVID-19 convalescence (define as at least 10 days after the onset of symptoms, no fever for at least 24 hours without the use of antipyretics and improvement of respiratory symptoms)
* informed consent signed
* clinical severity presentation of

  1. Severe the disease is classified as severe if one of the following conditions is met:

     Respiratory distress, respiratory rate ≥30/min Oxygen saturation on room air at rest ≤93%. Partial pressure of oxygen in arterial blood/FiO2 ≤300 mm Hg. Or
  2. Critical if one of the following conditions is met. Respiratory failure and mechanical ventilation are required. Shock occurs Another organ dysfunction is present
* risk of health complication >50% according to the health risk calculator
* less than 14 days of hospital discharge.

Exclusion Criteria:

* concomitant use of another anticoagulant
* known pregnancy
* known hypersensitivity to sulodexide
* need for hospital care at screening
* renal insufficiency with CrCl <30ml/min or continuous renal replacement therapy, hemodialysis, or peritoneal dialysis.
* blood platelet count < 30 000/µL
* other conditions that are judged to carry an increased risk of bleeding as judged by the Investigator
* more than 30 days of clinical onset

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2022-04-01 (Actual); Primary Completion 2022-09-01 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
Serum level of soluble Thrombomodulin | 8 weeks
  The level of serum soluble Thrombomodulin will be measured at 0, 4, and 8 weeks by ELISA test to detect endothelial dysfunction and its improvement.

SECONDARY OUTCOMES:
Serum level of Von Willebrand factor | 8 weeks
  The level of serum Von Willebrand factor will be measured at 0, and 8 weeks by ELISA test to detect pro-thrombotic status, endothelial dysfunction, and their improvement.
Serum level of ICAM-1 | 8 weeks
  The level of serum ICAM-1 will be measured at 0, and 8 weeks by ELISA test to detect pro-inflammatory status, endothelial dysfunction, and their improvement.
Serum level of VCAM-1 | 8 weeks
  The level of serum VCAM-1 will be measured at 0, and 8 weeks by ELISA test to detect pro-inflammatory status, endothelial dysfunction, and their improvement.
Serum level of soluble P-selectin | 8 weeks
  The level of serum soluble P-selectin will be measured at 0, and 8 weeks by ELISA test to detect pro-inflammatory status, pro-thrombotic changes, endothelial dysfunction, and their improvement.
Serum level of circulating endothelial cells | 8 weeks
  The level of circulating endothelial cells will be measured at 0, and 8 weeks by standardized flow cytometry to detect endothelial dysfunction and its improvement
Serum level of high sensitive C reactive protein | 8 weeks
  The level of high sensitive C reactive protein will be measured at 0, and 8 weeks by ELISA test to detect pro-inflammatory status, endothelial dysfunction, and their improvement.
Serum level of Interleukine-6 | 8 weeks
  The level of serum Interleukine-6 will be measured at 0, and 8 weeks by ELISA test to detect pro-inflammatory status, endothelial dysfunction, and their improvement.

OTHER OUTCOMES:
Serum level of D-dimer | 8 weeks
  The level of serum D-dimer will be measured at 0, 4, and 8 weeks by ELISA test to detect pro-inflammatory status, pro-thrombotic changes, endothelial dysfunction, and their improvement.
Serum level of fibrinogen | 8 weeks
  The level of serum fibrinogen will be measured at 0, 4, and 8 weeks by ELISA test to detect pro-inflammatory status, pro-thrombotic changes, endothelial dysfunction, and their improvement.
Platelets count in peripheral blood | 8 weeks
  Platelets count in peripheral blood will be measured at 0, 4, and 8 weeks by standard automatic analyzer for complete blood count to detect pro-inflammatory status, pro-thrombotic changes, endothelial dysfunction, and their improvement.
Post-COVID-19 functional status | 8 weeks
  Post-COVID-19 functional status will be assessed at 0, 4, and 8 weeks by a specific questionnaire "Post-COVID-19 Functional Status (PCFS)" scale that ranges from 0 (no limitations) to 4 (severe limitations).
Clinical progression of COVID-19 | 8 weeks
  Clinical progression of COVID-19 will be assessed at 0, 4, and 8 weeks by a specific World Health Organization Clinical progression scale that ranges from 0 (no infection) to 10 (death due to infection).
Thrombotic complications | 8 weeks
  Venous (deep vein thrombosis, superficial vein thrombosis, pulmonary embolism) and arterial (myocardial infarction, stroke, acute limb ischemia) thrombosis will be assessed on a clinical basis and should be confirmed by appropriate imaging (duplex ultrasound scan, computed tomography scan with contrast, arterial and venous angiography).
Major bleeding as defined by International Society on Thrombosis and Haemostasis (ISTH) criteria | 8 weeks
  Major bleeding as defined by the International Society on Thrombosis and Haemostasis (fatal bleeding, and/or symptomatic bleeding in a critical area or organ, such as intracranial, intraspinal, intraocular, retroperitoneal, intraarticular or pericardial, or intramuscular with compartment syndrome, and/or bleeding causing a fall in hemoglobin level of 2 g/dL (1.24 mmol/L) or more, or leading to transfusion of two or more units of whole blood or red cells) will be assessed on a clinical basis and should be confirmed by appropriate laboratory and instrumental tests.
Clinically relevant non-major bleedingas defined by International Society on Thrombosis and Haemostasis (ISTH) criteria | 8 weeks
  Clinically relevant non-major bleeding as defined by the International Society on Thrombosis and Haemostasis (requiring medical intervention by a healthcare professional, and/or leading to hospitalization, and/or increased level of care prompting a face to face [i.e., not just a telephone or electronic communication] evaluation) will be assessed on a clinical basis and should be confirmed by appropriate laboratory and instrumental tests.

CONTACTS AND LOCATIONS:
Overall Officials: Kirill Lobastov, PhD, Principal Investigator — Pirogov Russian National Research Medical University
Locations (1):
- Moscow Clinical Hospital no.24, Moscow, Russia

IPD SHARING:
Plan to Share IPD: No